CLINICAL TRIAL: NCT00193167
Title: Phase II Study of Weekly Topotecan in Patients Treated for Metastatic Colorectal Cancer
Brief Title: Weekly Topotecan in Patients Treated for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 56; 104864724
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
This non-randomized phase II study is designed to assess the response rate and toxicity of weekly topotecan as second-line treatment in patients with relapsed or refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Topotecan

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic colorectal cancer
* One previous chemotherapy for metastatic disease
* Measurable or evaluable disease
* Able to perform activities of daily living with assistance
* Adequate bone marrow, liver, and kidney function
* All patients must give written informed consent prior to study entry.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Brain or meningeal involvement
* Serious active infection or underlying medical conditions
* Other active neoplasms are ineligible
* Pregnant or lactating

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
overall response rate

SECONDARY OUTCOMES:
median survival
one year survival
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States